CLINICAL TRIAL: NCT06979843
Title: Evaluation of a Psychosocial Support Model for Adolescents and Young Adults Newly Diagnosed With Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Sophiahemmet University (Other); Vastra Gotaland Region (Other Government); Region Stockholm (Other Government)
Responsible Party: Principal Investigator, Jeanette Winterling, Associate professor, registered nurse, Region Stockholm
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Dnr 2024-07540-01
Record Dates: First submitted 2025-05-06; First posted 2025-05-20 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: The research design follows the framework for developing and evaluating complex interventions, applying a non-randomised design since the project aims at aligning as closely as possible to the clinical practice and everyday routine. Further, when an evidence-based intervention is implemented in another setting to wherein it was previously found to be effective, it is reasonable to evaluate both the intervention as well as the implementation process part. It is essential to include a process evaluation to be able to investigate aspects beyond effectiveness. A process evaluation can shed light on fidelity and quality of implementation, how is change produced and how is context affecting the implementation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- A psychosocial model (Experimental): The first aim is to evaluate if participating in the psychosocial model (including Team Young and PRISM) maintains or improves psychological resilience, psychological wellbeing, quality of life and hope among AYAs at a six-month follow-up, compared to time of diagnosis. The second aim is to evaluate how participants in the model of psychosocial support (including Team Young and PRISM) experience it with regard to acceptability, relevance and benefit.
  Interventions: Other: A psychosocial model

INTERVENTIONS:
Other: A psychosocial model — The first aim is to evaluate if participating in the psychosocial model (including Team Young and PRISM) maintains or improves psychological resilience, psychological wellbeing, quality of life and hope among AYAs at a six-month follow-up, compared to time of diagnosis. The second aim is to evaluate how participants in the model of psychosocial support (including Team Young and PRISM) experience it with regard to acceptability, relevance and benefit.
  The design is a longitudinal cohort study.

SUMMARY:
Rational:

Adolescents and young adults (AYAs) newly diagnosed with cancer is a small but vulnerable group with many psychosocial needs persisting for a long time. No standardized psychosocial support program exists for this group of patients in Sweden.

The program:

The program in the present project aims at offering all AYAs, newly diagnosed with cancer, at two Comprehensive Cancer Centres in Sweden, an individual information meeting with a "Team Young" to assess psychosocial needs and then offer available psychosocial support including a structured psychosocial program labelled Promoting Resilience in Stress Management (PRISM). PRISM aims to strengthen key resilience resources such as stress-management, goal setting, cognitive reframing, and meaning-making. It has been developed and evaluated in the US. Evaluations from the US have proven to be promising among AYAs with cancer. PRISM was associated with clinically and statistically significant improvements in resilience, hope, benefit-finding, disease-related quality of life, and reductions in psychological distress, compared to usual care. Our research group has translated and adopted PRISM to a Swedish context with a participatory research approach involving clinicians, researchers, and end-users. The first version of PRISM has been evaluated in a feasibility study and based on the findings revised. A second feasibility study was finalised during 2024 at two Comprehensive Cancer Centers in Sweden with preliminary findings indicating positive experiences from participants. In parallel to this project, comparison data on primary and secondary outcomes, has been collected from the general population in the same age group. The findings indicate so far promising psychometric properties for the main outcome resilience.

Aim:

The overall aim of this research project is to evaluate a psychosocial support program for adolescents and young adults (AYAs) newly diagnosed with cancer. It includes offering all AYAs, newly diagnosed with cancer, an information meeting with a "Team Young" to assess psychosocial needs and then offer available psychosocial support including a structured psychosocial program labelled Promoting Resilience in Stress Management (PRISM).

Method:

The design is a longitudinal cohort study and will include approximately 130 AYAs (16-30 years) newly diagnosed with cancer at Karolinska- and Sahlgrenska University Hospitals. All participants will complete questionnaires on three occasions: at enrolment in PRISM, after 4 modules in PRISM and six months after enrolment. The primary outcome measure is psychological resilience and secondary outcomes are psychological well-being, quality of life and level of hope.

Relevance:

Implementing a structured psychosocial support program for AYAs newly diagnosed with cancer has the potential to mean a lot for each patient and their families and facilitate for health care professionals involved in their cancer care.

If this research project shows promising results on resilience, psychological wellbeing, quality of life and/or hope, PRISM can be implemented as standard care at hospitals in Sweden treating AYAs with cancer.

ELIGIBILITY:
Inclusion Criteria for patients:

* Participants will be AYAs newly diagnosed with cancer at Karolinska University Hospital and Sahlgrenska University Hospital who have been referred to Team young by their contact nurse.
* Individuals newly diagnosed with cancer, 16-30 years of age who understand and speak Swedish.

Exclusion criteria for patients:

- Any psychiatric disorder or cognitive difficulties.

Inclusion criteria for health care professionals:

- Participants will be all eligible health care professionals, involved in delivering the implemented model of psychosocial support (Team Young and PRISM) at Karolinska University Hospital and Sahlgrenska University Hospital.

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 142 (Estimated)
Dates: Start 2025-01-16 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Resilience | Data collection implies all participants to complete questionnaires on three occasions: at enrolment in the study, after module 4 in PRISM (approximately 4-8 weeks after enrolment) and six months after enrolment in PRISM.
  The primary outcome, i.e. resilience will be measured with the Connor-Davidson Resilience Scale (CD-RISC-10 items). Score range is 0-40 for CD-RISC-10, with higher scores indicating greater resilience

CONTACTS AND LOCATIONS:
Overall Officials: Jeanette Winterling, Principal Investigator — Region Stockholm
Locations (2):
- Sweden (2):
  - Sahlgrenska University Hospital, Gothenburg
  - Karolinska University Hospital, Stockholm

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Odling M, Jervaeus A, Wengstrom Y, Rosenberg AR, Yi-Frazier JP, Winterling J. Adaptation and feasibility of the Swedish Promoting Resilience in Stress Management intervention targeting adolescents and young adults newly diagnosed with cancer. J Psychosoc Oncol. 2025;43(4):513-529. doi: 10.1080/07347332.2024.2419663. Epub 2024 Oct 28. PMID 39466132